CLINICAL TRIAL: NCT00210067
Title: A Double-Masked, Randomized, Dose-Ranging Study of a Single Intravitreal (IVT) Injection of INS37217 Intravitreal Injection in Subjects With Retinal Detachment
Brief Title: A Study in Subjects With Retinal Detachment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-101
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — denufosol tetrasodium; Intravitreal Injections

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Intravitreal Injection

SUMMARY:
The purpose of this trial is to access the tolerability of INS37217 Intravitreal Injection when administered intravitreally in subjects with macula-on or macula-off rhegmatogenous retinal detachment (RRD).

ELIGIBILITY:
Inclusion Criteria:

* have macula-on or macula-off rhegmatogenous retinal detachment
* are eligible for pneumatic retinopexy, with identifiable retinal breaks
* are phakic or pseudo-phakic

Exclusion Criteria:

* have detachments not of a rhegmatogenous nature
* currently have blood in the vitreous, corneal opacity, or other conditions which limit the view of peripheral retina
* have evidence of intraocular inflammation (uveitis)
* have a history of current condition of uncontrollable, elevated IOP or open-angle glaucoma
* have breaks not conducive to a single procedure of pneumatic retinopexy treatment
* have proliferative vitreoretinopathy of type C or D
* have previously had a vitrectomy or require one
* have previously had a scleral buckle procedure

Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-05; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
tolerability

SECONDARY OUTCOMES:
pharmacological activity

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director